CLINICAL TRIAL: NCT04028674
Title: Functional Electrical Stimulation of the Bilaterally Paralyzed Human Larynx
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, David Zealear, PhD, Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 200932; 5U01DC016033-05 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bilateral Vocal Fold Paralysis (BVFP)

STUDY DESIGN:
Intervention Model Description: Following implantation of the laryngeal pacing device and post-operative visit, participants will be randomized to their treatment group (Early Activation vs. Delayed Activation) and unilateral stimulation side (Right PCA vs. Left PCA) using the REDCap randomization module.
  1. To treatment group at a 1:1 ratio-Either the Early Activation Group (n=4) or the Delayed Activation Group (n=4)
  2. To unilateral stimulation side at a 1:1 ratio-The side for unilateral stimulation will be either the left PCA muscle (n=4), or the right PCA muscle (n=4)
Who Masked: Outcomes Assessor
Masking Description: The blinded procedures include PIF, CAPE-V, NGA, X-Tol.
  * PIF: A research staff member will be unblinded and control the pacer programmer. The testing condition will be programmed prior to start of test. Both patient and staff administering the test will be blinded to testing condition.
  * CAPE-V: Clinically-certified SLPs involved in perceptual ratings of voice quality will be blinded to experimental testing condition and data collection timepoint.
  * NGA: NGA is analyzed from stills of the glottis collected during endoscopy. These images will be randomized and de-identified before analysis to blind the rater.
  * X-Tol: A research staff member will be unblinded and control the pacer programmer. The testing condition will be programmed prior to start of test. Both patient and staff administering the test will be blinded to testing condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Early Activation of Laryngeal Pacing device (Experimental): Early Activation of the laryngeal pacing device (n=4) at one-month post-implantation.
  Interventions: Device: Laryngeal Pacing Device
- Delayed Activation of Laryngeal Pacing device (Sham Comparator): Delayed activation of the laryngeal pacing device (n=4) at two months post-implantation.
  Interventions: Device: Laryngeal Pacing Device

INTERVENTIONS:
Device: Laryngeal Pacing Device — Device is an implantable neurostimulation system designed to deliver low-intensity electrical impulses to nerve structures.

SUMMARY:
The primary purpose of this project is to evaluate the safety of new treatment termed bilateral laryngeal pacing to improve treatment outcomes in patients with bilateral vocal fold paralysis (BVFP) (Aim 1). Outcome measures related to voice and ventilation will also provide initial insights into the efficacy of bilateral (Aim 2) and unilateral (Aim 3) stimulation of the implanted device to improve treatment outcomes in patients with BVFP.

DETAILED DESCRIPTION:
Despite recent advances in medicine, rehabilitation of the paralyzed larynx remains a complex clinical problem. Based on national health statistics, it is anticipated approximately 7,000 patients will be diagnosed with BVFP in the United States each year. BVFP is a serious and often life-threatening clinical condition. The recurrent laryngeal nerve (RLN) carries motor fibers that innervate both the abductor muscle (posterior cricoarytenoid muscle) and adductor muscles of the vocal folds. Damage to the nerve compromises both of these functions and arrests the vocal folds in a near-closed position. With BVFP, voice tends to be functional, but airway compromise is often severe enough to warrant tracheotomy to relieve inspiratory stridor and dyspnea. If spontaneous recovery does not occur within one year, it is likely that the patient's vocal folds will be chronically paralyzed. In such instances, long-term tracheostomy can be considered. Unfortunately, permanent tracheostomy is associated with complications such as tracheal stenosis, chronic infection, and psycho-social impairment. For this reason, laryngeal surgery is usually recommended to enlarge the airway and restore breathing through the mouth. Procedures such as arytenoidectomy, cordotomy, or repeated Botox injections, regarded as the standard of care for enlarging the airway, also have inherent complications. Specifically, they impair voice and compromise airway protection during swallowing. The limitations associated with these current treatments have prompted investigation into a more physiologic, dynamic approach to rehabilitation: reanimation of the paralyzed PCA muscle by functional electrical stimulation (FES). Ideally, stimulation should be applied during the inspiratory phase of respiration to abduct the vocal folds. This has been termed "laryngeal pacing". During non-inspiratory phases, stimulation would cease, and the vocal folds would passively relax to the midline to allow for normal voice production and airway protection. Previously, our clinical trial of unilateral pacing demonstrated a significantly greater return of ventilation without any compromise of voice or swallowing. However, the level of ventilation was only marginally better than that associated with cordotomy.

In the current project, we will investigate the safety of a novel intervention (laryngeal pacing) for BVFP (Aim 1). The overarching hypothesis is that neuromuscular activation of the PCA muscles bilaterally reestablishes bilateral glottal opening and ventilation through the mouth without alteration of voice or swallowing, compared to a sham-operated control (Aim 2). The ventilation from bilateral pacing should be significantly greater than from unilateral pacing and allow the patient to engage in a normal pre-paralysis activity level (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Willingness to comply with all study procedures and availability for the duration of the study.
* Male or female adult patients, 22 years of age or older.
* Diagnosis of one of the following at least ten months prior to study enrollment:

  * Complete bilateral vocal fold paralysis, with suspected etiological event occurring at least ten months prior to study enrollment. Diagnosis will be documented via medical records and confirmed during the onsite screening visit by a Vanderbilt board certified laryngologist via endoscopy, electromyography and direct laryngoscopy.
  * Incomplete bilateral vocal fold paralysis (severe paresis) which significantly impedes respiration may also be considered for participation under the same conditions and per physician recommendation. Patients must present with an NGA less than 20, representing severe laryngeal obstruction. Diagnosis will be documented via medical records and confirmed during the onsite screening visit by a Vanderbilt board certified laryngologist via endoscopy, electromyography, and direct laryngoscopy.
* Patients receiving repeated botulinum toxin (botox) injections into the thyroarytenoid muscle to treat BVFP may be eligible for participation per physician recommendation.
* Demonstrated glottal opening bilaterally (abductory response) upon percutaneous needle stimulation of PCA muscles (i.e. mean NGA ≥0.05 per vocal fold tested).
* Patients who have previously undergone a recurrent laryngeal nerve reinnervation procedure may be eligible for participation per physician recommendation. Patients must have undergone the laryngeal nerve reinnervation surgery at least 10 months prior to enrollment in the laryngeal pacing study.
* Patients who have previously undergone a recurrent laryngeal nerve reinnervation procedure may be eligible for participation per physician recommendation. Patients must have undergone the laryngeal nerve reinnervation surgery at least 10 months prior to enrollment in the laryngeal pacing study.
* Patients with or without a tracheostomy
* Demonstrated glottal opening bilaterally (abductory response) upon percutaneous needle stimulation of PCA muscles (i.e. mean NGA ≥0.05 per vocal fold tested).

Exclusion Criteria:

* Any active illness that is associated with an auto-immune disorder (such as diabetes).
* History of cardiac dysrhythmias or implanted cardiac pacemaker.
* Cardiac irregularities identified in screening electrocardiogram.
* Any electronic implanted medical device that, in the investigator's opinion, could interact with the laryngeal pacemaker.
* Active cardiac disease manifested by unstable angina, recent myocardial infarction, malignant arrhythmias, uncontrolled hypertension (diastolic greater than 110), or decompensated congestive heart failure.
* Patients with underlying comorbidities that, in the investigator's opinion, could potentially warrant a need for oxygen therapy, including but not limited to: Chronic obstructive pulmonary disease, asthma, emphysema, recurrent bronchitis, pneumonia or interstitial lung disease.
* Bilateral laryngeal immobility from stenosis or arthritis.
* Poor surgical risk patients as determined by the treating surgeon or Vanderbilt Preoperative Evaluation Center (VPEC).
* The abundance of interstitial fat may impede the surgical dissection. In the opinion of the principal investigator or treating physician(s), patients with factors that may complicate the surgical intervention will be excluded.
* Known allergy to barium dye or anesthetics.
* Known allergy to any of the device materials.
* History of aspiration pneumonia, secondary to bilateral vocal fold paralysis
* Persistent thin liquid dysphagia despite standard of care dysphagia management strategies (e.g. small sips, chin tuck, etc.)
* Presence of significant tracheal narrowing.
* Any anatomical abnormality that would jeopardize safe implantation, per the surgeon.
* Any medical condition, that in the opinion of the principal investigator or treating physician would jeopardize the outcome or welfare of the participant.
* Any previous medical treatment that in the opinion of the principal investigator or treating physician would confound the effects of laryngeal pacing.
* Females who are pregnant or plan a pregnancy within 2 years. A pregnancy test will be done as part of the routine pre-operative assessment for all females of child-bearing potential.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improved ventilation due to laryngeal pacing device as assessed by increase in standard assessment testing (peak inspiratory flow or PIF). | 12 months
Better voice quality as assessed by decrease in standard assessment testing (Consensus Auditory Perceptual Evaluation of Voice or CAPE-V). | 12 months

SECONDARY OUTCOMES:
Increased glottal area due to laryngeal pacing device as assessed by increase in normalized glottal area (NGA) results. | 12 months
Increase in exercise tolerance due to laryngeal pacing device as assessed by treadmill testing. | 12 months
Better quality of life (QOL) outcomes due to laryngeal pacing device, self assessed via patient reported outcome surveys. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David L. Zealear, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No